## **SUMMARY OF CHANGES**

# **ANCHOR Study: Anal Cancer Prevention Study**

Anal Cancer/HSIL Outcomes Research Study Version 15.0

NCI Protocol #: AMC-A01 Local Protocol #: ANCHOR

NCI Version Date: 22JAN2021 Protocol Date: 22JAN2021

# I. Scientific and Substantive Changes

| # | Section | Description of Change |
|---|---|---|
| 1. | Additional Studies, Health- Related Quality of Life Study, Attachment 1 | The ICF was revised to implement the A-HRSI instrument as a formal QoL aim, among participants who opt in to complete this questionnaire. The questionnaire will be given to up to 500 participants in English or Spanish at 8 time points. Participants will be paid \$25 for each completed time point. |
| 2. | Additional Studies, Oral and Anal COVID Infection | The ICF was revised to add an optional study for investigating SARS-CoV-2 in oropharyngeal and anal swab samples from PLWH being screened for the ANCHOR study at 2 time points. Participation is limited to 5 centers: Laser Surgery Care, Anal Dysplasia Clinic MidWest, University of Miami (including Jackson Memorial Hospital), Grady Memorial Hospital, and University of California, San Francisco; centers not participating in this substudy must not offer this optional study in the local informed consent form. Participants will be paid \$10 for each completed time point. |
| 3. | Are there any payments? | Information shared with ClinCard was updated to remove protected health information (SSN) that is not added to the system. |

# II. Administrative and Editorial Changes

| # | Section | Description of Change |
|---|---|---|
| 4. | <u>Footer</u> | The footer was updated to version 15.0, dated 22JAN2021. |
| 5. | Who will see my medical information? | The manufacturer name for topical medications was updated from Valeant Pharmaceuticals to Bausch Health. |

### MODEL INFORMED CONSENT FORM

**Study Title for Study Participants:** 

ANCHOR: Anal Cancer Prevention Study

Official Study Title for Internet Search on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>:

ANCHOR: Anal Cancer/HSIL Outcomes Research Study

# What is the usual approach to preventing anal cancer?

You are being asked to take part in this study because you are an adult with HIV infection and you may have anal high-grade squamous intraepithelial lesions (HSIL). Anal HSIL is tissue in the anal canal that has been damaged by human papillomavirus (HPV) and is at risk for turning into anal cancer.

There is no standard approach for preventing anal cancer. Some doctors try to prevent anal cancer by looking for and treating anal HSIL. The treatments may vary.

# What are my other choices if I do not take part in this study?

If you decide not to take part in this study, you have other choices. For example:

- You may choose not to be screened or treated for anal HSIL.
- You may choose to be screened or treated for anal HSIL outside of this study.

# Why is this study being done?

This goal of this study is to see whether treating anal HSIL will prevent anal cancer compared with watching HSIL carefully without treatment (active monitoring). We will compare the number of people who develop anal cancer in both groups. We know that treating HSIL in the cervix can prevent cervical cancer in women. However, we don't know if treating anal HSIL can prevent anal cancer. For this reason, most doctors in the United States don't look for and treat anal HSIL. Anal cancer is more common in women and men with HIV than in the general population. If caught early, anal cancer is often cured, but treatment-related side effects can be severe and some can last for several years. Anal HSIL occurs before cancer develops and is quite common in HIV-infected people (between 10% and 50% have anal HSIL). Most cases of anal HSIL will never become cancer.

# What are the study groups?

5,085 men and women will take part in this study. To be in the study, you need to be 35 years of age or older, have HIV infection, have not been treated for anal HSIL in the last 6 months, and have never had cancer of the anus, vulva, vagina, or cervix. If you have anal HSIL and you meet the other eligibility criteria, you can join this study. A computer will assign you by chance (like tossing a coin) to join one of the two study groups: Active Monitoring (Group 1) or Treatment (Group 2). This is called randomization. You have an equal chance (50/50) of being assigned to either group. We do not know if one group is better than the other and that is why you are being assigned to one of the groups.

• Group 1 (Active Monitoring) will not have any HSIL treatment

• Group 2 (Treatment) will have treatment of anal HSIL chosen by you and your study provider

Another way to find out what will happen to you during this study is to read the chart below. Start reading at the left side and read across to the right, following the lines and arrows.



# What are the advantages of being in Group 1 or Group 2?

The researchers estimate (an educated guess) that the risk of developing anal cancer if your HSIL is not being treated is about 1 in 100 over the course of the study.

## **Advantages to Group 1 (Active Monitoring)**

• Treating anal HSIL may not be better than active monitoring to reduce the risk of anal cancer, and if so, you would have avoided uncomfortable treatments that provide little benefit to you.

## **Advantages to Group 2 (Treatment)**

• If you are in the treatment arm your HSIL may be reduced in size or removed entirely.

# How long will I be in this study?

The researchers plan to recruit volunteers for the study over a period of three years or more. We will follow all participants for up to five years after the last participant joins the study. Participants who join the study in the first year may be in the study for up to eight years or more. If anal cancer is found at any time during the study, your participation in the study will end, and you will be immediately referred for the necessary treatment. If at any time during the study, the results show that treatment is helpful in preventing anal cancer, and you still have anal HSIL, you will be referred for treatment.

# What extra tests and procedures will I have if I take part in this study?

• Most of the exams, tests, and procedures you will have are part of the usual approach for anal HSIL among those doctors who routinely choose to screen and treat this disease. Samples collected only for experimental laboratory research studies are shown in **bold.** All research samples are required for this study. The samples will be tested at the end of the study for different factors related to HPV, anal HSIL and anal cancer. The results of the research tests will not be given to you or your doctor.

## **Before you begin the study:**

- You will take a brief questionnaire (<u>Attachment 3</u>) to be sure the information in this consent form is clear. The questionnaire will take about five minutes to complete.
- You will have a screening visit. During this visit, we will ask you about your medical history and perform tests to confirm that you can be in this study. We will ask you to bring in your HIV medication(s). You should avoid receptive anal intercourse, enemas, or inserting anything in your anus for 24 hours before all study visits.
- A physical exam including a genital exam.
- Three anal swabs. The researcher will put a swab (similar to a Q-tip<sup>TM</sup>) into your anus. The end of the swab will be rubbed against the skin inside the anus. This swab is for anal cytology (Pap test) to test for abnormal cells in the anus. The leftover cells from the first swab, and all of the cells from the second and third swabs are for future research studies.
- An anal/rectal exam with a finger.
- An anal exam called high resolution anoscopy (HRA) that uses a special microscope to find abnormal areas of the anus. A lubricated plastic anoscope will be inserted into your anus. Then, a piece of gauze moistened with acetic acid (i.e., vinegar) is placed in your anus so that abnormal areas will show up. The researcher puts the anoscope back into your anus. A colposcope (a machine with a magnifying lens) is used to see the skin inside the anus. Iodine may be used to help make lesions show up.
- Anal biopsies: These are pieces of anal skin about the size of a sesame seed that are cut out to look for HSIL under a microscope. Your provider may inject a small amount of local anesthesia (numbing medicine) before the biopsy. Your biopsy may be re-read by another doctor at another institution to check your diagnosis. If the provider finds anal cancer, we will ask you to return to the clinic for an extra anal biopsy for future research studies before you stop the study.
- **Blood** will be drawn (about 4 teaspoons) to check your blood cell counts, to test for HIV unless we have a copy of your HIV test results, and **for future research studies**.
- A pregnancy test, if you are a woman who could become pregnant.

If you are not eligible for the study, with your permission, we may use the information and samples that we have collected for future research. If you are eligible then you will be randomized at your next visit to Group 1 (Active Monitoring) or Group 2 (Treatment). A study calendar that shows what will be done during the study for both groups is attached.

# For all participants who enroll in the study:

- We will ask about your medical history and sexual behaviors at your Visit 1
- At each 6-month visit you will have three anal swabs for anal cytology and **future research studies**
- Digital anal/rectal exam, and HRA
- Depending on which group you are in, you may or may not have one or more anal biopsies at any one visit. A part of your biopsies may also be used for future research studies.

- 1½-3 teaspoons of blood will be collected for future research studies
- We will call you between visits to ask about any side effects from study procedures, answer questions about the study, and what the study team can do to make future study visits easier.

If the provider finds anal cancer at any visit, we will ask you to return to the clinic for an extra anal biopsy for future research studies before you stop the study.

## **If you are in Group 1 (Active Monitoring):**

- You will have biopsies of your anal HSIL every year. Your provider may choose to perform biopsies every 6 months or see you in between 6-month visits at any time if there is any concern that cancer has developed.
- It is important that you do not receive any other treatment for anal HPV-related disease outside of this study. If you have anal warts and want to have them treated, the study doctors will treat them and you may continue in the study.
- If at any time during the study, the results show that treatment is helpful in preventing anal cancer, and you still have anal HSIL, you will be referred for treatment.

## If you are in Group 2 (Treatment):

- The study doctor will talk to you about your treatment options for HSIL. Please see the attachment for the description of treatments available in this study and the follow-up required for each of these treatments. You will receive treatment as soon as you start the study.
- You may have additional visits after treatments to watch for any side effects and extra biopsies to see how the treatment is working. You will have biopsies at least once per year and probably more often.
- Participants receiving some of the treatments in the clinician's office may have **one additional biopsy for future research studies** every 6 months, just before getting treatment.
- During the study, the study doctor may try different treatments if your HSIL does not go away or comes back.

## **Treatments used in the Treatment Arm include:**

- Imiquimod 5% cream, which is also known as Aldara<sup>™</sup>. This treatment is an approved treatment of genital warts (skin growths caused by HPV). You apply this cream yourself to the inside or outside of your anus, depending on where your HSIL is found.
- Topical 5-fluorouracil (5FU) cream, also known as Efudex<sup>TM</sup>. 5FU cream is approved for treating actinic keratosis (precancerous conditions of the skin not related to HPV), and for superficial basal cell carcinoma (a skin cancer not related to HPV). You apply this cream yourself to the inside or outside of your anus, depending on where your HSIL is found.
- Imiquimod and 5FU are experimental when used to treat anal HSIL.
- Infrared coagulation, or IRC, which is a method that uses a device to destroy or remove a specific area of skin using a focused beam of light. IRC is approved for treating anal warts and removing tattoos. It is experimental for treating anal HSIL.

- Electrocautery, also known as hyfrecation, involves the use of an electric probe that is used to destroy or remove a specific area of skin. A laser may also be used. These are approved by the FDA for use in surgical procedures.
- Surgery in the operating room to cut out the HSIL (this is an uncommon approach (less than 10% of the time) and is only used if none of the other treatments can be used.

# What possible risks can I expect from taking part in this study?

If you choose to take part in this study, there is a risk that:

- You may lose time at work or home and spend more time in the hospital or doctor's office than usual.
- You may be uncomfortable being asked sensitive or private questions
- The study treatments for anal HSIL may not be better, and could possibly be worse, than doing nothing for your anal HSIL.
- The researchers estimate (an educated guess) that the risk of developing anal cancer if your HSIL is not being treated is about 1 in 100 over the course of the study. We do not know what the risk is among those whose anal HSIL is being treated.

<u>Anal swabs for cytology and research material</u>: Putting a swab into the anus may cause some discomfort. Minor bleeding (less than a quarter of a teaspoon) occurs in some people due to the insertion of the swabs. The bleeding stops almost right away.

<u>High resolution anoscopy</u>: Insertion of an anoscope will likely cause some discomfort. You may feel pressure and the urge to have a bowel movement. Putting acetic acid (vinegar) in the anal canal may cause minor burning and irritation.

<u>Anal biopsies</u>: You may have pain with the anal biopsies. You may have some bleeding for up to a week after biopsies, especially when you have a bowel movement. There is a rare chance of very heavy bleeding that may require extra treatment. There is a very slight risk of infection (<1%). Contact the study clinic if you have symptoms of heavy bleeding or infection (fever, pain, redness, or swelling).

<u>Local anesthetic</u> (numbing medicine): You may have a pinching or burning feeling from the shot of numbing medicine. There is a very slight chance of reaction to the numbing medicine including rash, flushing, rapid heartbeat, and dizziness.

<u>Blood drawing (venipuncture) risks</u>: In many people, obtaining blood from a vein may cause some discomfort. This may include infection, bruising, and/or tenderness at the site where the blood is taken, and fainting or feeling faint.

<u>Questionnaire</u>: You will be asked questions about any sex you have had recently. Some people may find these questions embarrassing. It is important that you answer these questions honestly. However, no one will force you to answer any questions if it is too uncomfortable for you.

## Additional risks for those in Study Group 1 – Active Monitoring

#### COMMON

You may be anxious if you are concerned that your HSIL may progress to cancer and you are not undergoing active treatment

## Additional risks for those in Study Group 2- Treatment

In addition to the side effects outlined above, people in Group 2 may also experience the possible side effects of the study treatments received. The tables below show the most common and the most serious side effects that researchers know about for each agent. There might be other side effects that researchers do not yet know about. If important new side effects are found, the study doctor will discuss these with you.

## Risks of topical imiguimod 5%

### COMMON, MILD TO MODERATE

In 100 people receiving imiquimod, more than 20 and up to 100 may have:

- Pain, burning, irritation, and itching
- Redness
- Swelling
- Ulcerations (i.e., sores on the skin) and bleeding
- Flaking and crusting of the skin
- Allergic reactions near treatment area
- Pain, redness and sores on skin near the treatment area (for example on the scrotum in men)

## OCCASIONAL, MILD TO MODERATE

Of 100 people receiving imiquimod, from 4 to 20 may have:

- Headache
- Rash at other sites
- Back pain
- Sinus infection, nausea, fever, and flu-like illness

### RARE, AND SERIOUS

Of 100 people receiving imiquimod, 3 or fewer may have:

• The common skin reactions described above may be severe enough that your study provider may stop the medication for a while or try a lower dose of the medication. You may also need other treatments such as pain medications to treat this.

## Risks of topical 5-fluorouracil 5% (5-FU)

### COMMON, MILD TO MODERATE

Of 100 people receiving 5FU, more than 20 and up to 100 may have:

- Pain, burning, irritation and itching
- Redness
- Swelling
- Ulcerations (i.e., sores on the skin) and bleeding
- Flaking and crusting of the skin
- Allergic reactions in the skin
- Pain, redness and sores on skin near the treatment area (for example on the scrotum in men)
- Scarring of the skin

## OCCASIONAL, MILD TO MODERATE

Of 100 people receiving 5FU, from 4 to 20 may have:

- Emotional upset, trouble sleeping, irritability
- Medicinal taste in your mouth
- Low platelet counts, high white blood cells counts, and other blood count problems.
- Loss of hair, and other rashes.
- Red irritated eyes, and irritated nose
- If you have had herpes infection in the past, it may cause it to return.

## RARE, AND SERIOUS

Of 100 people receiving 5FU, 3 or fewer may have:

- Extensive skin reactions. The common skin reactions described above may be severe enough that your study provider may stop the medication for a while or try a lower dose of the medication. You may also need other treatments such as pain medications to treat this.
- There have been miscarriages (loss of a pregnancy), and one birth defect (a serious heart condition) in women who have used 5FU during pregnancy.

## Risks of infrared coagulation (IRC), laser, and electrocautery

### COMMON, MILD TO MODERATE

Of 100 people receiving IRC/electrocautery/laser, 50 or more may have:

- Slight pain during the treatment
- Some spotting or drops of blood on toilet tissue paper for up to 2 weeks after the treatment.
- Mild to moderate pain that may continue for up to 2 weeks after the treatment, usually well controlled with pain or anti-inflammatory medicines. There may be a change in the texture of the treated area for 1 to 2 weeks.

### RARE, SOME MAY BE SERIOUS

Of 100 people receiving IRC/electrocautery/laser, 1 or fewer may have:

- Fistula formation (a tunnel between two skin surfaces)
- Severe bleeding (typically 7-10 days after the procedure) which may need additional treatment
- Abscess (an infection under the skin resulting from the procedure)
- Scarring, which could keep stool from passing normally
- Pain that is severe and lasts longer than 2 weeks.

Additional risks: If you have had herpes infection in the past, the treatment may cause it to return.

## Risks of surgical excision (cutting out the lesion), or treatment under anesthesia

## **COMMON, SOME MAY BE SERIOUS**

Of 100 people receiving treatment under anesthesia, from 50 or more may have:

- Bleeding after the procedure
- Pain, sometimes severe for up to 2 weeks after the procedure
- Difficulty having a bowel movement

## OCCASIONAL, SOME MAY BE SERIOUS

Of 100 people receiving treatment under anesthesia, fewer than 20 may have:

• Changes in the coloring (more pigment or darkening, or less darkening) of their skin when treated for disease on the outside of the anus

### RARE, SOME MAY BE SERIOUS

Of 100 people receiving treatment under anesthesia, 1 or fewer may have:

- Abscess (an infection under the skin resulting from the procedure)
- A tear or hole in the anus or rectum that may require surgery
- A bad reaction to the anesthesia, up to and including death
- Scarring, which could keep stool from passing normally

If you have a biopsy or are treated with IRC, electrocautery, laser, or surgery, you should not have receptive anal sex for up to 2 weeks after treatment. This is to allow you to heal. You may have some bleeding with receptive anal sex until healing is complete.

If you are selected to participate in Group 2 (Treatment arm), you may need more than one kind of treatment to treat your HSIL over the course of the study. It is possible that the doctors may not be able to remove all of the HSIL. It is possible that anal HSIL treatment may not prevent cancer.

Reproductive risks: The study drugs used in this study could be very damaging to an unborn baby.

- Female participants should not get pregnant while in this study. Women who could get pregnant should use at least one form of birth control during the study and for 3 months after stopping all study treatment.
- Male participants should not father a baby while receiving topical study drugs (creams). Men who could father a child should use at least one form of birth control during treatment with topical study drugs and for 2 weeks after stopping all treatment.

Check with the study doctor about what types of birth control, or pregnancy prevention, to use while in this study. Please tell the study doctor immediately if you become pregnant or if your partner becomes pregnant during this study. If you get treatment with 5-FU or imiquimod, your partner should wear a condom if you have receptive anal sex to avoid exposure to these drugs.

## *Here are important points about side effects:*

- The study doctors do not know who will or will not have side effects.
- Some side effects may go away soon, some may last a long time, or some may never go away.

Here are important points about how you and the study doctor can make side effects less of a problem:

- Tell the study doctor if you notice or feel anything different so they can see if you are having a side effect.
- The study doctor may be able to treat some side effects.
- The study doctor may adjust the study drugs to try to reduce side effects.

Let your study doctor know of any questions you have about possible side effects. You can ask the study doctor questions about side effects at any time.

# What possible benefits can I expect from taking part in this study?

It is not possible to know at this time if treating anal HSIL is better than the usual approach (not treating it) in reducing the risk of anal cancer so this study may or may not help you. This study will help researchers learn which approaches could help people in the future.

# Can I stop taking part in this study?

Yes. You can decide to stop at any time. If you decide to stop for any reason, it is important to let the study doctor know as soon as possible so you can stop safely. We would like you to continue in the study even if you decide to stop HSIL treatments or undergoing study procedures. If you agree to stay in the study but cannot come to the clinic, we will contact you once a year until the study is over to ask whether you were diagnosed with anal cancer. The study doctor will tell you about new information or changes in the study that may affect your health or your willingness to continue in the study.

The study doctor may take you out of the study:

- If your health changes and taking part in the study is no longer in your best interest.
- If new information becomes available.
- If you do not follow the study rules.
- If the study is stopped by the sponsor, Institutional Review Board (IRB), National Cancer Institute (NCI), or the Food and Drug Administration (FDA).

# What are my rights in this study?

Taking part in this study is your choice. No matter what decision you make, and even if your decision changes, there will be no penalty to you. You will not lose medical care or any legal rights.

# What are the costs of taking part in this study?

Your health plan/insurance company will need to pay for all of the standard costs of treating or watching your anal HSIL while in this study. This includes the cost of study tests (high resolution anoscopy, anal cytology (Pap smear)), and anal biopsies, the costs of the study treatments, and the cost of any medicines needed to manage any side effects. At the screening visit, if your health insurance plan will not cover these costs, the study will pay for your HRA, anal biopsies, and anal cytology at screening. Neither you nor your insurance company will pay for any of the research specimens or tests. Before you decide to be in the study, you should check with your health plan or insurance company to find out exactly what they will pay for, and what you may be personally responsible for in the form of a co-pay or deductible. The study may be able to reimburse you for any out-of-pocket costs that you may have for study visits, including copays and deductibles. You should discuss this with the study staff to see if you are eligible for reimbursement for these expenses, including what paperwork and documents you will need to provide. If you and/or your

health insurer are unable to pay for the associated standard of care costs, you can meet with a financial counselor to determine if you are eligible for the research to cover these costs. If you do not have insurance, then all costs related to study procedures, visits, and laboratory tests will be covered by the study. The study cannot cover any costs for medical care outside of study visits. If the study ends early, the study will not be able to continue to cover the costs of your care.

# Are there any payments for taking part in this study?

You will not be paid for taking part in this study. However, the study will reimburse you \$100 for your time and expenses for every scheduled study visit where HRA is performed. You will be reimbursed \$25 for study visits where only swabs are collected. Also, you may receive a small thank-you gift when you reach a milestone in the study, such as a one-year visit. (Instruction to site: modify as required for local limits on participant payments. Add any additional retention incentives or gifts based as required by local IRB policy).

(Omit paragraph if site is not using ClinCard for reimbursement) You will receive reimbursement for this study using a "ClinCard." ClinCard is managed by a company called Greenphire. ClinCard works like a prepaid credit card and can be used where MasterCard is accepted. At a minimum, your name, initials, and date of birth will be given to Greenphire to load funds on your ClinCard. If you agree, you may also provide your email and/or cell phone number to Greenphire to receive email or text notifications when funds are loaded to your ClinCard. If you sign up for text reminders, you may be charged by your cell phone carrier for the texts, depending on your plan. Greenphire will not be given any of your medical information. Let the research staff know if you have concerns about using ClinCard.

The study staff will do everything possible to make your visits as easy as possible and may provide additional assistance with transportation and childcare.

# What happens if I am injured or hurt because I took part in this study?

If you are injured or hurt as a result of taking part in this study and need medical treatment, please tell your study doctor. The study sponsors will not offer to pay for medical treatment for injury. Your insurance company may not be willing to pay for study-related injury. If you have no insurance, you would be responsible for any costs.

If you feel this injury was a result of medical error, you keep all your legal rights to receive payment for this even though you are in a study.

# Who will see my medical information?

Your privacy is very important to us and the researchers will make every effort to protect it. Your information may be given out if required by law. For example, certain states require doctors to report to health boards if they find a disease like gonorrhea. However, the researchers will do their best to make sure that any information that is released will not identify you. Some of your health information, and/or information about your specimen, from this study will be kept in a central database for research. Your name or contact information will not be put in the database.

There are organizations that may inspect your records. These organizations are required to make sure your information is kept private, unless required by law to provide information. Some of these organizations are:

- The University of California, San Francisco, and the AIDS Malignancy Consortium (AMC), the organizations that are conducting this study
- The Institutional Review Board, IRB, is a group of people who review the research with the goal of protecting the people who take part in the study
- The Food and Drug Administration and the National Cancer Institute
- The pharmaceutical collaborator, Bausch Health, and other companies who provide support for the study
- The AIDS and Cancer Specimen Resource at the University of Arizona, the specimen bank for the ANCHOR Study
- If you request to be seen at a new ANCHOR Study site, we will share your study records with the new ANCHOR site

## Where can I get more information?

You may visit the NCI Web site at http://cancer.gov/ for more information about studies or general information about cancer. You may also call the NCI Cancer Information Service to get the same information at: 1-800-4-CANCER (1-800-422-6237).

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# Who can answer my questions about this study?

| You can talk to the study doctor a | bout any questions or concern | s you have about this study or to |
|---|---|---|
| report side effects or injuries. Cont | act the study doctor | (insert name of study |
| doctor[s]) at | _ (insert telephone number). | |

## **Additional Studies Section**

This section is about optional studies you can choose to take part in:

## **Optional Donation of Leftover Tissue Samples**

After all of the tests for the ANCHOR study are finished, there may be unused blood, anal swab, and biopsy tissue left over. We would like your consent to donate your leftover samples for future research studies. If you agree, your samples will be stored in the AIDS and Cancer Specimen Resource (ACSR). The ACSR is funded by the National Cancer Institute (NCI) to collect, store, and distribute samples from research study participants to qualified scientists. This research may be about cancers and pre-cancers associated with HIV disease. This future research will be approved by the study researchers and the NCI.

Donating your leftover samples will not require any extra tests or procedures. You are free to choose if you want to donate your leftover samples. You do not have to donate your leftover samples to take part in this study. If you do not give your consent, we will destroy your leftover samples at the end of the study.

The researchers will send the ACSR some medical information from your study records. This information may be useful to researchers who perform studies using your samples. The researchers will not give the ACSR your name or any information that could personally identify you. The

researchers will make every effort to protect your privacy. The ACSR will label your samples with codes and store them for future testing.

You may withdraw your samples from the ACSR at any time. You may contact the study coordinator if you would like to withdraw your samples. The coordinator can ask in writing that your sample be removed from research use and that any identifiable sample and information still in their possession be destroyed. However, if any research has already been done using some of your samples, the data will be kept and analyzed as part of those studies.

You may not have any direct benefit from donating your leftover samples to the ACSR. However, research done using your samples may help other people in the future. These studies may help us learn more about how to prevent and treat HIV-associated cancers. You will not be paid for donating your leftover samples to the ACSR.

# **Genetic Testing**

Some of your samples may be used for genetic testing to understand how anal HSIL progresses to anal cancer. Someone might be able to trace this information back to you. While the ACSR and researchers who study your samples for any genetic testing will have no information that could identify you, there is a risk that someone could use information from genetic studies to trace your samples back to you. The researchers believe the chance that someone will identify you is very small, but the risk may change in the future as people come up with new ways of tracing information. In some cases, this information could be used to make it harder for you to get or keep a job. There are laws against misuse of genetic information, but they may not give full protection. None of the results of any genetic tests done with your samples will be reported back to you or the study doctor.

You may contact the research team if you have any questions about donating your leftover samples.

## Anal Health-Related Symptom Index (A-HRSI) Quality of Life Questionnaire

You may choose to participate in optional questionnaires to measure how monitoring or treating your anal HSIL in this study affects your quality of life. This study is being run with researchers at Memorial Sloan Kettering Cancer Center (MSKCC). This study involves taking the A-HRSI questionnaire with twenty-five questions at eight different times, asking you to rate symptoms of your HSIL. These questions ask about such things as pain, problems moving, and enjoyment of sexual activity. The A-HRSI questionnaire may only be taken in English or Spanish. Up to 500 participants may take part.

You may take the questionnaire using a computer, tablet, or smartphone without going to the clinic. You will be asked to provide your phone number to take part in this study. If you do not have a phone but want to take part, you can go to the clinic to take the questionnaire over the phone.

If you agree to take part and if you are eligible to be in the ANCHOR Study, you will take the A-HRSI questionnaire once before you are randomized in the main study, and at 7 other times after randomization (2-7 days, 4 weeks, and 12, 24, 36, 48, and 60 months after randomization). After each questionnaire, we will ask you to confirm your phone number and email for reminders, how you want to take the questionnaire next time, and if you want to get text or email reminder messages for the next questionnaire.

If you agree to get reminder messages, we will also collect the name of your cell phone carrier and email address to send you text or email reminders to take the questionnaires. This contact

information will be shared with ANCHOR Study staff at The Emmes Company to send you these reminder messages. The study team at the clinic will also use your contact information for reminder calls, to help you access the electronic questionnaire, or to ask you to complete it over the phone. The research team will not share your contact information with any other parties.

Answering the questions should take about 6-10 minutes each time. There is a risk you may be embarrassed by the questions asked. You will not receive any direct benefits from this study. It will help the researchers measure how treating or watching anal HSIL affects patients' quality of life. If you wish to stop participating, you may do so at any time.

If you do not wish to take the questionnaire on a computer you may complete the questionnaire by phone. If you take the questionnaire by phone, you will use some of your data or minutes on your phone plan, and may risk running out. If you do not have a phone, or do not wish to use your phone for this study, you may complete the questionnaire at the site on a computer or using a site phone. If you have a change in phone number or phone carrier, you will need to contact the study team to let them know.

Participants will be paid \$25 for each of the eight times that they take the A-HRSI questionnaire (\$200 total). This payment will be made using your ClinCard. [Site to specify method of payment if different from ClinCard.]

You may contact the research team if you have any questions about participating in the quality of life questionnaire.

### SARS-CoV-2 (COVID-19) oral and anal infection

(Note to sites: only the 5 participating ANCHOR sites may include this section in the local informed consent form)

We would like your consent to take part in an optional study to research how often PLWH have oral and/or anal infection with SARS-CoV-2, the virus that causes COVID-19. We will also study if there is any relationship between SARS-CoV-2 and anal HPV infection. Lastly, we will study if SARS-CoV-2 infection has any effect on anal HSIL or anal HPV persisting or going away. Up to 400 participants will take part in this optional study.

If you agree, we will collect an oropharyngeal swab (a swab of the back of the throat, like a swab to test for strep throat) before you start the study. If you are enrolled into the study, we will collect another oral swab at visit 2 (6 months). This must be done at the same visit that anal swab samples are collected. We will use a portion of your anal swab samples from the Biorepository from these two visits for this study. Everyone who comes to an ANCHOR Study site for a study visit is asked about symptoms or possible exposure to COVID-19 and if you are participating in this optional COVID-19 study, we may use that information in our study analysis.

These samples will be sent to UCSF for testing. You will not get the results of your tests since they will not be run until the end of this substudy and will not be used for your medical care. If you think you have COVID-19 symptoms or have been exposed to someone with COVID-19, please talk to a healthcare provider immediately to make sure that you get the necessary medical care.

You are free to choose if you want to take part in this substudy. If you agree to take part and we collect your samples, but your screening evaluations show that you are not eligible for ANCHOR, you can still take part in this study. Any samples we have collected will still be used for this study.

You may withdraw your samples from this substudy at any time. You may contact your study coordinator if you would like to withdraw your samples. The coordinator can ask in writing that your sample be removed from research use and that any identifiable sample and information be destroyed. However, if any research has already been done using some of your samples, the data will be kept and analyzed as part of this study.

There are no costs to take part in this substudy. You will receive \$10 via your ClinCard at the visits where oral swabs are collected for participating in this optional study.

You may not have any direct benefit from participating in this optional study. However, research done using your samples may help other people with COVID-19 and/or anal HSIL and anal HPV in the future.

# **Samples for Future Research Studies**

If I am enrolled in the ANCHOR study, my leftover samples and related information may be donated to the ACSR for use in future health research. (circle one)

YES NO

I agree to have my samples undergo genetic testing to learn about, prevent, diagnose, or treat HIV-related diseases and cancer. (circle one)

YES NO

# **Research Use of Your Screening Visit Samples**

If I am ineligible for the study, or choose not to participate in the study, the researchers may use my study data and samples collected during the screening visit for future research. (circle one)

YES NO

## **Future Studies**

We may want to call you in the future to see if you may be interested in being in other studies.

If you are called, you can decide if you want to be in any of the other studies and would sign another form to be in those studies. You are free to decide whether or not you want us to call you. Your decision about being called later for other studies will not change your being in this study.

The researchers may call me about taking part in future studies. (circle one)

YES NO

# Anal Health-Related Symptom Index (A-HRSI) Quality of Life Questionnaire

I agree to participate in the A-HRSI questionnaires. I understand that I need to provide a phone number or go to the clinic to participate in this substudy. I acknowledge that clinic staff will contact me to complete the questionnaires over the phone if I do not take the questionnaires at the site or online (circle one).

YES NO

If yes, I prefer to complete questionnaires (circle one)

ONLINE BY MYSELF SITE STAFF CALLS ME AT THIS CLINIC

If yes, I prefer to complete questionnaires (circle one)

| IN ENGLISH IN SPANISH | |
|---|---|
| My preferred phone number for clinic staff to contact me for this study is: | |
| I agree to receive email reminders for taking ques<br>if you agree to these reminders) | tionnaires (circle yes and provide email address |
| YES TO EMAIL REMINDERS | NO EMAIL REMINDERS |
| Email address (for sending computer-generated en | nail reminders): |
| I agree to receive text message reminders for taken phone information if you agree to these reminders | · , |
| YES TO TEXT REMINDERS | NO TEXT REMINDERS |
| Cell phone number (check here if number is the sa | ame as preferred phone number above): |
| Cell phone carrier name (for sending computer-ge | enerated text message reminders): |
| CONTACT BETWEEN STUDY VISTS (option agreement) | nal, include only if site has a Mosio business |
| This ANCHOR study site would like to send you to ANCHOR appointments and to check in with you letexts is optional and you can request that we stop contract with Mosio.com, a secure, HIPAA-compressages and act on your responses to them. As a messages will be able to see our message. If you asked to provide a cell phone number to rece coordinator. If you sign up for text reminders, you the texts, depending on your plan. | between ANCHOR study visits. Receiving these sending you reminders at any time. We have a cliant texting service to help us send these text reminder, anyone with access to your phone text consent to receive these messages, you will be ive text messages from the ANCHOR study |
| I agree to be contacted via text message for the Al | NCHOR study (circle one) |
| YES NO | |
| My preferred cell phone number for receiving text | ts from this ANCHOR site is: |

# **SARS-CoV-2 Optional Study**

| (Note to sites: only the 5 participating AN informed consent form) | NCHOR sites may include this section in the local |
|---|---|
| I agree to take part in the optional SARS-Co | V-2 study. (circle one) |
| YES NO | |
| This is the end of the section about additional | l research studies. |
| My Signature Agreeing to Take Par | t in the Main Study |
| | o me. I have discussed it with the study doctor and my en a signed copy of this form. I agree to take part in here I circled 'yes'. |
| Participant's Signature | Date of Signature |
| Signature of Person(s) conducting the Informed Consent Discussion | Date of Signature |

# **Attachment 1: ANCHOR: Anal Cancer Prevention Study**

# **Group 1 Study Calendar for Participants, Active Monitoring**

The list below describes the required study visits and the tests and procedures that will be done for each visit on the Active Monitoring Arm (Group 1). The researchers will not perform any study procedures unless you give your consent to take part and the tests and procedures from the screening visit show that you can take part in the study.

## VISIT 1 (Month 0) – Baseline Visit, Enrollment, Randomization (1-12 weeks after screening)

- Review of any signs or symptoms or changes in your medications.
- The anal health-related quality of life questionnaire (A-HRSI), if you agreed to take this survey. This questionnaire asks about how your anal HSIL symptoms affect you. It takes less than 10 minutes to complete.
- The ANCHOR Visit 1 Questionnaire, which asks questions about your smoking history, drug use, sexual history, and medical conditions and diagnoses related to anal disease. This questionnaire will take approximately 25 minutes to complete.
- Blood sample for HIV viral load and CD4 count.
- Urine pregnancy test if you are a woman who could become pregnant.
- An anal exam with a gloved finger and a groin exam for lumps or tenderness.
- High resolution anoscopy.
- The study team will tell you your randomization assignment. The procedures below are only for participants assigned to Group 1, the Active Monitoring arm.
- After visit 1, and all other study visits, a member of the study team will call you to remind you of your next visit. The study staff will ask if there is anything that the study team can do to make it easier for you to attend the study visits. (Note: insert information on local activities and support for retention if relevant to the site)
- If you agreed to take the A-HRSI questionnaire, you will take it home on the internet or by phone call at 2-7 days and 4 weeks after Visit 1. See the information sheet on the A-HRSI for more instructions.

# VISITS 2, 4, 6, 8, and 10 – Six-Month Visits (Months 6, 18, 30, 42, 54, and later visits after Month 60 as required)

- Review of any signs or symptoms or changes in your medications.
- Questions about your HIV viral load and CD4 count from routine medical care.
- Physical exam, including vital signs.
- Anal swab for anal cytology and research.
- Two more anal swabs for **research**.
- An anal exam with a gloved finger and a groin exam for lumps or tenderness.

- High resolution anoscopy. The study doctor will only collect anal biopsies at this visit if there are any areas that show signs of getting worse or progressing to cancer. A part of your biopsies may also be used for **research studies**.
- Blood sample for research studies.

# VISITS 3, 5, 7, 9, and 11 – Annual Visits (Months 12, 24, 36, 48, 60, and later visits after Month 60 as required)

- All of the items listed above. In addition you will have biopsies of all anal HSIL lesions.
- If the provider finds anal cancer at any visit, we will ask you to return to the clinic for an extra anal biopsy for future research studies before you stop the study.
- If you agreed to take the A-HRSI questionnaire, you will take it at month 12, 24, 36, 48, and 60.

## Final Study Visit (Month 60 or later)

- You will have all of the evaluations listed above.
- You will have biopsies of all anal HSIL lesions and areas that used to have HSIL but now appear to be normal. If this totals less than 4 biopsies, normal-appearing tissue will be biopsied so that at least 4 areas are sampled.
- If you still have anal HSIL after the final study visit is complete, the researchers will contact you. You will be referred for appropriate medical care outside of this study.

# **ANCHOR: Anal Cancer Prevention Study**

# **Group 2 Study Calendar for Participants, Treatment**

The list below describes the required study visits and the tests and procedures that will be done for each visit on the Treatment Arm (Group 2). The researchers will not perform any study procedures unless you give your consent to take part and the tests and procedures from the screening visit show that you can take part in the study.

## VISIT 1 (Month 0) – Baseline Visit, Enrollment, Randomization (1-12 weeks after screening)

- Review of any signs or symptoms or changes in your medications.
- The anal health-related quality of life questionnaire (A-HRSI), if you agreed to take this survey. This questionnaire asks about how your anal HSIL symptoms affect you. It takes less than 10 minutes to complete.
- The ANCHOR Visit 1 Questionnaire, which asks questions about your smoking history, drug use, sexual history, and medical conditions and diagnoses related to anal disease. This questionnaire will take approximately 25 minutes to complete.
- Blood sample for HIV viral load and CD4 count.
- Urine pregnancy test if you are a woman who could become pregnant.
- An anal exam with a gloved finger and a groin exam for lumps or tenderness.
- High resolution anoscopy.
- The study team will tell you your randomization assignment. The procedures below are only for participants assigned to Group 2 (the Treatment arm).
- The study doctor will show you how to apply any topical treatments, or will perform or schedule your first treatment for anal HSIL.
  - o Imiquimod 5% cream: you will insert the cream inside or outside your anus, depending on where the HSIL was found, with a gloved finger three times per week for up to 16 weeks.
  - o 5% FU cream: you will apply the cream inside or outside your anus, depending on where the HSIL was found, with a gloved finger twice per day for five days, then take a break from treatment for 9 days (14 day cycle). You will have up to 8 of these 14-day treatment cycles (up to 16 weeks total).
  - o Infrared coagulation (IRC), hyfrecation/electrocautery, or laser ablation: during an HRA exam, the study doctor will apply the treatment tip of the medical device to your HSIL lesion. Before this treatment, the researcher will inject the lesions with a local anesthetic (lidocaine or other anesthetic). You may have **one additional biopsy for future research studies** every 6 months, just before getting treatment. You may have multiple treatments on any given lesion that will last for a second or two each. Any dead tissue from the treatment will be cut away from the treatment site. The researcher may also treat other HPV lesions such as anal warts with the device. You may have repeat treatments within the next 8 weeks depending on the amount of disease.

- O Surgery to remove HSIL (treatment under anesthesia): If the study doctor believes that none of the treatment approaches above will help to get rid of HSIL, you will be referred to a surgeon and will have surgery with anesthesia to remove the HSIL. You may have repeat procedures after 8 or 12 weeks for follow-up if the HSIL is still present. This treatment will only be recommended as a last option.
- After Visit 1, and all other study visits, a member of the study team will call you to remind you of your next visit. The study staff will ask if there is anything that the study team can do to make it easier for you to attend the study visits. (Note: insert information on local activities and support for retention if relevant to the site.)
- If you agreed to take the A-HRSI questionnaire, you will take it home on the internet or by phone call at 2-7 days and 4 weeks after Visit 1. See the information sheet on the A-HRSI for more instructions.

# Visits 1A and IB – Interim Treatment Visits for Imiquimod 5% or 5-FU (8 weeks, and possibly 16 weeks after Visit 1)

- At 8 weeks, you will have Visit 1A
  - o Review your signs and symptoms and any changes to your medications.
  - o An anal exam with a gloved finger and a groin exam for lumps or tenderness.
  - o High resolution anoscopy exam to see how you are responding to treatment.
  - o If you are a woman who could become pregnant, you will have a urine pregnancy test.
- If the study doctor recommends that you continue treatment for 8 more weeks, you may be asked to return at 16 weeks (Visit 1B) for another follow-up visit with the same procedures listed above.
- You may have one additional biopsy every 6 months for research purposes.

# Visit 1A – Interim IRC, Electrocautery, or Laser Ablation Treatment Visits (up to 8 weeks after Visit 1)

- Within 8 weeks after randomization, you will have Visit 1A
  - o Review your signs and symptoms and any changes to your medications.
  - o An anal exam with a gloved finger and a groin exam for lumps or tenderness.
  - o High resolution anoscopy exam to see how you are responding to treatment.
  - o If you are a woman who could become pregnant, you will have a urine pregnancy test.
  - o If the study doctor recommends that you continue treatment, or there are more lesions to treat, you will have another ablation treatment at this visit.

# VISITS 2-10+ – Six-Month Visits (Months 6, 12, 18, 24, 30, 36, 42, 48, 54, and later visits after Month 60 visits as required)

- Review of any signs or symptoms or changes in your medications.
- Questions about your HIV viral load and CD4 count from routine medical care.
- Physical exam, including vital signs.

- Anal swab for anal cytology and research.
- Two additional anal swabs for **research**.
- An anal exam with a gloved finger and a groin exam for lumps or tenderness.
- Blood sample for research studies.
- If you are a woman who could become pregnant, you will have a urine pregnancy test before getting any treatments.
- High resolution anoscopy. The study doctor will collect biopsies of any lesions that look like HSIL. A part of your biopsies may also be used for **research studies**.
- You will receive your next study treatment if needed or discuss treatment changes with the study doctor.
- If you agreed to take the A-HRSI questionnaire, you will take it at month 12, 24, 36, 48, and 60.
- You will have additional visits for treatment follow-up after each 6-month visit when treatment is given (e.g., Visit 2A, 2B for imiquimod treatment), as described above under Visit 1.
- If the provider finds anal cancer at any visit, we will ask you to return to the clinic for **an extra** anal biopsy for future research studies before you stop the study.

## Final Study Visit (Month 60 or later)

- You will have all of the evaluations listed above.
- High resolution anoscopy. You will have biopsies of all anal HSIL lesions. If no lesions are seen, the study doctor will take biopsies of areas that were treated to be sure that there is no more anal HSIL. If this totals less than 4 biopsies, normal-appearing tissue will be biopsied so that at least 4 areas are sampled.
- If you still have anal HSIL after the final study visit is complete, the researchers will contact you. You will be referred for appropriate medical care outside of this study.

# **Attachment 2: Diagram of the Anus**



# **Attachment 3: ANCHOR Study Comprehension Assessment**

Instructions: We would like to ask you some questions about the ANCHOR Study to be sure that the information we provided about study was clear. Please read each statement about the ANCHOR Study below. Please circle the best response or "I don't know" if you do not know the answer.

| Name: | Date: |
|------------------------------------|-------|
| 1. Once I sign the consent form, I | |

- a. can never leave the study.
- b. must provide a compelling reason for leaving the study.
- c. can only leave the study after consulting with the study investigators.
- d. can leave the study at anytime for any reason.
- e. I don't know.

### 2. What is HPV?

- a. cancerous tissue.
- b. a procedure where a clinician will insert a scope into the anus.
- c. a virus that can potentially cause anal cancer.
- d. a wart.
- e. I don't know.
- 3. What are high grade squamous intraepithelial lesions (HSIL)?
  - a. areas of skin damaged by HPV.
  - b. cancerous tumors.
  - c. anal warts that turn white with vinegar.
  - d. a sexually transmitted infection.
  - e. I don't know
- 4. Why is this study being done?
  - a. To find a cure for HPV.
  - b. To find a cure for HIV.
  - c. To find out if anal cancer is caused by HIV and HPV infection.
  - d. To find out if treating HSIL prevents anal cancer.
  - e. I don't know

- 5. How long will I be followed if I enroll in the study?
  - a. 1-2 years
  - b. 3-4 years
  - c. 5-8 years
  - d. for as long as I have HSIL
  - e. I don't know
- 6. If I am in the active monitoring group, what is expected of me?
  - a. I will not have to come in for visits.
  - b. I will be given a cream, surgery, or heat/laser to remove my HSIL.
  - c. I will come in for visits every 6 months but will not have any anal biopsies.
  - d. I will come in for visits every 6 months, will have biopsies at least every year, and my HSIL will be closely monitored by the clinician.
  - e. I don't know.
- 7. If I am in the treatment arm, what is expected of me:
  - a. I will not have to come in for visits.
  - b. I will come in for visits every 6 months but will not have any anal biopsies.
  - c. All of the treatments will take place in the operating room.
  - d. I may undergo several courses of treatment, and possibly different kinds of treatment, over the course of the study.
  - e. I don't know.
- 8. Can I switch from the study group to which I have been assigned to the other study group:
  - a. No, I can't switch to the other study group at any time during the study.
  - b. Yes, I can switch to the other study group within the first year after I join the study.
  - c. Yes, I can switch to the other study group at any time during the study.
  - d. Yes I can switch to the other group and then switch back if I want to.
  - e. I don't know.

Informed Consent Instructions for Study Staff (omit from local ICF document given to study participants):

Administer the questionnaire to the participant after the informed consent discussion has occurred before the participant signs the informed consent form. After the participant provides responses, review the answers to the questionnaire with the participant, and re-review or provide additional information as relevant to all incorrect responses to answer any questions. If the participant declines to answer any questions, the correct responses may be reviewed with the participant. There is no minimum score requirement for the assessment; follow-up to the questionnaire is important to reinforce key information about the study and assist comprehension before the participant provides consent to participate. The completed Attachment 3 and documentation of the research staff's review of this assessment with the participant must be maintained in the site's source documents with the participant's signed informed consent form for all screened participants.

## Answer Kev

- 1. D
- 2. C
- 3. A
- 4. D
- 5. C
- 6. D
- 7. D
- 8. A

# **Attachment 4: ANCHOR Informed Consent Frequently Asked Questions**

#### What is HPV?

- "Human papillomavirus" is a virus passed between people during sex
- Some of the 80 different types of HPV cause warts, while others can cause cancer, including cervical or anal cancer
- HIV weakens the immune system and reduces the body's ability to fight HPV, increasing the risk of warts and cancer

### What is HSIL?

- "High-grade squamous intraepithelial lesions"
- HSIL is tissue damaged by 1 or more types of HPV
- This tissue is at risk of turning into cancer
- HSIL is common among people living with HIV

#### Is HSIL anal cancer?

- No, HSIL is pre-cancer, HSIL rarely becomes cancer
- We estimate that 1 in 100 HIV+ people with HSIL will develop anal cancer after 5 years

# How is HSIL treated and what are the risks of treatment?

- HSIL can be removed with one or more laser, heat or acid treatments, a daily cream, or surgery
- Treatment side effects can be severe, but for laser, heat or acid treatments only last a short time, usually less than a week; Side effects due to the cream may last longer

### Why is this study being done?

We don't know if treating HSIL prevents anal cancer

### Who can be in the study?

- We need 5,085 people to volunteer for 5-8 years
- 35 years of age or older
- Living with HIV (we'll need to see which meds you're on)
- Have not been treated for anal HSIL in the last 6 months
- Never had anal, vulvar, vaginal, or cervical cancer
- Must have anal HSIL found during screening

### What possible benefits can I expect in this study?

- You may not benefit from the study, because we don't know what's best: treatment or monitoring
- This study will hopefully benefit future generations

### What happens in the study?

- Volunteers receive either treatment or monitoring
- After 5-8 years, we will compare cancer rates by group

### Can I choose which study group I am in?

- No a computer randomly assigns you
- Once you're in your group, that's your group

### Other than this study, what are my choices?

Manage HSIL outside of this study

### What are the advantages of being in each group?

- Active Monitoring: Treating anal HSIL may not be better than active monitoring to reduce the risk of anal cancer. If so, you would have avoided uncomfortable treatments that provide little benefit to you.
- Treatment: If you are in the treatment arm your HSIL may be reduced in size or removed entirely.

### What tests and procedures happen in both groups?

- Physical/genital exam: 1st visit & maybe more often
- 3 anal swabs: every 6 months
- Finger exam: every 6 months
- Anoscopy (also called HRA): every 6 months, maybe more often
- Biopsies: once per year, maybe more often
- Blood draw: every 6 months
- Pregnancy test: at screening and before treatments
- Follow-up phone call: every 6 months

### What are the general risks in this study?

- Screening and treatment procedures may cause discomfort; please see full consent for details
- You may lose work time while recuperating

### Are all of these tests and procedures necessary?

- Two anal swabs, blood samples, and some anal biopsies are extra
- These will be kept for future research

### What happens to my leftover tissue after the study?

- You can donate these for future studies
- Some samples may be used for genetic testing
- You can say no to donating your samples and still be in the ANCHOR study

### What's expected of me in "active monitoring"?

- Study visits every 6 months
- More frequent visits if cancer is suspected

### How long will I be in the study?

5 to 8 years or longer, with your permission

### What's expected of me in "treatment"?

- HSIL treatment in consultation with a study doctor
- Possibly extra visits & biopsies to check for side effects and to see if treatment has removed HSIL
- If HSIL doesn't go away/returns, more treatment
- Women should not get pregnant while they are in the study
- Men who could father a baby should use birth control (condoms) while using topical creams to treat HSIL

#### What are the treatment side effects?

- Each treatment has common side effects
- Some treatment side effects can be severe
- Please see the full consent for details
- Always tell our doctor about your side effects; we can usually help you feel more comfortable

#### What are the specific risks of treatment?

The risks of your specific treatment will be discussed with you by your health provider.

#### Can I still have anal sex?

- Yes! but you will need time to heal for 2 weeks or more after procedures
- While using creams, sex partners should use a condom to avoid exposure to the chemicals

### What happens if I develop anal cancer?

The study stops for you and we refer you to cancer care

### Could the study end early?

Yes – if we learn that one group is better or that neither group is better at preventing anal cancer

#### Can I stop being in the study?

- Yes you may leave, at any time for any reason
- Always let our doctor know, so you can stop safely
- We'd like to stay in touch even if you stop visiting us

# Could my participation end earlier for other reasons?

- Yes if you cannot follow the study procedures
- Yes if the doctor takes you out of the study
- Yes if the study is stopped for administrative reasons
- Treat anal HPV/warts only with your study doctor

## • Biopsies (every year, possibly more often)

### What are my rights in this study?

- There's no penalty if you choose not to be in the study; you will not lose medical care or legal rights
- Questions? Call the IRB at [Phone]
- Email the IRB at [IRB email]

### What are my costs in this study?

- A co-pay or deductible, based on insurance coverage
- If you have no insurance, the study covers the costs

### Will I be paid for this study?

- No but we'll reimburse for your time and expenses as listed below
- When HRA is performed, we give you \$100
- When only swabs are taken, we give you \$25

### What if I'm hurt because of this study?

- If you're hurt or injured, please tell the study doctor
- You're responsible for medical treatment for injury
- You keep your legal rights to seek payment

### Who will see my medical information?

- We make every effort to protect your information
- Names and contact information are stored by local site and separately from ANCHOR clinical database
- Some organizations may inspect your records; they are required to keep your information private

### Where can I get more information about this study?

- 1-800-4-CANCER or http://cancer.gov
- http://www.clinicaltrials.gov/NCT02135419
- https://anchorstudy.org/

### Who can answer my questions about this study?

Contact [Site PI's name and phone number]

### Will the study interfere with my other healthcare?

- Generally speaking, your healthcare won't change
- But please treat HPV, including warts, only with us

### What should I do if I feel a change in my body?

- You know how your body feels, better than anybody
- A change in your body may be important
- Please tell our doctor, so we can pay attention too!

# **Attachment 5: Certificate of Confidentiality Statement**

# **ANCHOR: Anal Cancer Prevention Study**

Anal Cancer/HSIL Outcomes Research Study Conducted by the AIDS Malignancy Consortium (AMC)

The NIH has given the AMC and the ANCHOR Study researchers a Certificate of Confidentiality. The Certificate does not mean that the NIH or the U.S. Government recommend that you take part in this study. This Certificate helps us keep your health information private.

Your records for this study will have information that may identify you. This Certificate lets us turn down legal demands for your study records. We can use the Certificate to turn down demands for records from a U.S. court. The Certificate can be used in any federal, state, or local legal matters. We will use the Certificate to turn down any demands for your study records. The cases where we cannot use the Certificate are explained below.

We cannot use the Certificate to turn down a demand from the U.S. Government for study records. This applies to audits or reviews of the ANCHOR Study, or records that we have to report to the NIH or FDA.

The Certificate does not stop you or your family members from sharing your health information. It does not stop you from talking about taking part in this study. You may give written permission for an insurer, employer, or other person to get copies of your study records. If you give permission, we cannot use the Certificate to say no to a request for your study records.